CLINICAL TRIAL: NCT07160985
Title: AI-Assisted Blood Glucose Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Li Huating (Other)
Responsible Party: Sponsor-Investigator, Li Huating, Professor, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-06
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- X Life Lifestyle Guidance (Experimental)
  Interventions: Other: AI-based Lifestyle Management
- Standard Care (Active Comparator)
  Interventions: Other: Lifestyle Management

INTERVENTIONS:
Other: AI-based Lifestyle Management — Participants will use the X Life system for 28 days, receiving real-time, personalized dietary and exercise recommendations triggered by glucose level and activity tracker data. Participants can interact with the system by uploading meal images, physical activity data, and wearable-derived metrics.
  Arms: X Life Lifestyle Guidance
Other: Lifestyle Management — Participants will receive guideline-based lifestyle counseling according to national prediabetes prevention guidelines, delivered via mobile terminal, without AI-generated recommendations.
  Arms: Standard Care

SUMMARY:
AI-driven health management tools can leverage continuous glucose monitoring (CGM), physical activity, and dietary data to provide real-time, individualized feedback, improving self-management and adherence. The X Life model integrates AI algorithms with wearable devices to dynamically adjust dietary and exercise recommendations. Preliminary user studies suggest good usability and user experience, with potential to promote positive behavior change.

This trial aims to preliminarily evaluate whether the X Life AI system can improve glucose tolerance (measured by oral glucose tolerance test [OGTT] incremental area under the curve [iAUC]) in adults with prediabetes, providing effect size and protocol design reference for a future confirmatory randomized controlled trial. The investigators designed this trial with the assistance of a digital twin-based clinical research system (termed X Town).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Prediabetes (per ADA or WHO criteria)
* Stable lifestyle and body weight (±5%) for ≥3 months
* Owns and can operate a smartphone
* Able to understand and sign informed consent

Exclusion Criteria:

* Current glucose-lowering medication use
* Severe cardiovascular disease, liver/kidney dysfunction, or active malignancy
* Psychiatric or cognitive disorders affecting participation
* Planned major surgery or long-distance travel during the study
* Allergy/intolerance to CGM sensor materials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2025-09-07 (Actual); Primary Completion 2025-11-23 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in OGTT Glucose Incremental Area Under the Curve (iAUC) | Baseline and at the end of the 28-day intervention period.
  Difference between groups in the incremental area under the curve for plasma glucose concentration during a 2-hour oral glucose tolerance test (OGTT), calculated from measurements at 0, 60, and 120 minutes, adjusting for baseline values.

SECONDARY OUTCOMES:
Change in OGTT Plasma Glucose Levels | Baseline and at the end of the 28-day intervention period.
  Difference between groups in plasma glucose levels at 0, 60, and 120 minutes during OGTT, adjusting for baseline values.
Change in Continuous Glucose Monitoring (CGM) Metrics | Baseline (7-day run-in period) and during the 28-day intervention period.
  Difference between groups in CGM-derived metrics, including mean glucose, daytime TIR, nighttime TIR, glucose standard deviation (SD), coefficient of variation (CV), time above range (TAR >10.0 mmol/L), and time below range (TBR <3.9 mmol/L and <3.0 mmol/L).
Change in OGTT Plasma Insulin Levels | Baseline and at the end of the 28-day intervention period.
  Difference between groups in plasma insulin concentrations at 0, 60, and 120 minutes during OGTT, adjusting for baseline values.
Composite Body Composition Outcomes | Baseline and at the end of the 28-day intervention period.
  Body composition will be assessed and each measurement will be reported separately: Body weight, BMI (calculated from weight and height), Body fat percentage, Fat-free mass, Waist circumference, Hip circumference, Thigh circumference, Blood pressure (systolic and diastolic, reported separately).
Composite Metabolic Parameters | Baseline and at the end of the 28-day intervention period.
  Metabolic outcomes will be assessed and each laboratory parameter will be reported separately: Blood lipids: Total cholesterol, LDL-C, HDL-C, triglycerides; Liver function tests: ALT, AST, GGT; Kidney function tests: Serum creatinine, eGFR, etc.
Composite Patient-Reported Outcomes | Baseline, at the end of the 28-day intervention period and at the end of the 7-day follow-up period.
  Patient-reported outcomes will be assessed using validated questionnaires. Each scale will be reported and analyzed separately: WHO-5 Well-being Index: 0-25, higher = better well-being; Self-Efficacy: 10 items, each rated 1-4. Total score range 10-40; higher scores indicate stronger self-efficacy, etc.
User Experience Score with the X Life Model | At the end of the 28-day intervention period.
  User experience will be assessed using a questionnaire covering Knowledge & Awareness, Acceptability, Usability, Motivations & Barriers, Perceived Benefits and Perceived Risks. Each item is rated on a 5-point Likert scale. Higher scores indicate better user experience.
Safety and Tolerability | From baseline to the end of the 28-day intervention period.
  Incidence and frequency of adverse events (AEs), serious adverse events (SAEs), symptomatic and asymptomatic hypoglycemia (<3.9 mmol/L and <3.0 mmol/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China